CLINICAL TRIAL: NCT04495816
Title: COVID-19 Anosmia Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Alfred-Marc Iloreta, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 20-1132
Record Dates: First submitted 2020-07-30; First posted 2020-08-03 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Anosmia; Covid19
Keywords: Novel Coronavirus; Anosmia; Smell Loss; Parosmia; Fish Oil Supplement; Omega-3 Fatty Acid Supplements
MeSH Terms: conditions — Anosmia; COVID-19; Olfaction Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into treatment and control groups. The treatment group will receive omega-3-fatty acid supplementation (1000 mg of omega-3 fatty acid blend including 683 mg Eicosapentaenoic Acid and 252 mg Docosahexaenoic Acid) to be taken twice daily for 6 weeks. The control arm will receive a placebo pill to be taken twice daily.
Who Masked: Participant, Investigator
Masking Description: The healthcare providers interacting with the patients, as well as the participants themselves, will not know which arm they have been assigned to. Only the research fellows will have access to the randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 (Active Comparator): 1,000 mg of omega-3 fatty acid (2 softgels per day for 6 weeks)
  Interventions: Drug: Omega-3 Fatty Acid Supplement
- Placebo/Control (Sham Comparator): 2 softgels per day for 6 weeks
  Interventions: Drug: Placebo/Control

INTERVENTIONS:
Drug: Omega-3 Fatty Acid Supplement — Participants randomized to this arm will be instructed to take two of the softgels they received per day for 6 weeks. They will receive softgels containing 1,000 mg of omega-3 fatty acid. 1000 mg of omega-3 fatty acid blend including 683 mg Eicosapentaenoic Acid and 252 mg Docosahexaenoic Acid
  Arms: Omega-3
Drug: Placebo/Control — Patients randomized to this arm will also be instructed to take two of the softgels they received per day for 6 weeks. They will receive placebo softgels that are indistinguishable from those containing fish oil.
  Arms: Placebo/Control

SUMMARY:
To capture the natural history of COVID-19 associated olfactory dysfunction as measured by two patient reported outcome measures (SNOT-22, QOD-NS) and a 6-week BSIT with a comparison to an intervention arm receiving daily omega-3 supplements.

DETAILED DESCRIPTION:
Infection with the novel coronavirus (COVID-19) has been linked to new-onset olfactory dysfunction, often as the only presenting symptom. In one multicenter European study, 85.6% of patients with mild to moderate symptoms reported hyposmia or anosmia with early recovery of olfactory function in just under half of patients. However, the pathogenesis and natural history of COVID-19 related olfactory dysfunction is poorly understood.

Anosmia most commonly arises in association with sinonasal disease or post-infectious or post-traumatic disorders. Notably, olfactory loss has been associated with impaired quality of life, higher rates of depression, and even increased mortality risk. Spontaneous recovery has been observed in patients with post- infectious olfactory dysfunction, typically over a period of months to years, with an estimated one-third of patients demonstrating meaningful improvement after one year.

Smell retraining therapy appears to be an effective therapeutic option for patients with post-infectious olfactory dysfunction, particularly for patients who initiate treatment within one year from onset of symptoms, but requires an intervention period of at least three to four months. Various pharmacotherapies have been investigated in the treatment of post-infectious anosmia but none have clearly demonstrated utility with the exception of a possible benefit for nasal steroid irrigations in combination with smell retraining therapy.

More recently, omega-3 polyunsaturated fat supplementation has emerged as a promising pharmacotherapy for olfactory dysfunction in patients without sinonasal disease. Omega-3 fatty acid deficient mice demonstrate evidence of olfactory dysfunction and mice receiving omega-3 fatty acids have improved recovery after peripheral nerve injury, which has been linked to neuroprotective effects mediated through anti-oxidant and anti-inflammatory pathways. In humans, a large cross-sectional study found that older adults with higher dietary fat intake had lower incidence of olfactory impairment. From a clinical perspective, patients without sinonasal disease receiving postoperative omega-3 fatty acid supplementation after endoscopic endonasal skull base surgery in a randomized control trial demonstrated a significantly greater rate of return of normal olfactory dysfunction.

Little is known about either the natural history of olfactory dysfunction associated with COVID-19 infection or about the therapeutic efficacy of omega-3 fatty acid supplementation in patients with post-viral anosmia. The study team hopes to gain a better understanding of each through a randomized double-blind placebo control study that assesses both objective and subjective perception of olfactory dysfunction over a period of 6 weeks after infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older) with self-reported new-onset olfactory dysfunction
* Positive COVID-19 diagnosis will be deemed eligible for inclusion.

Exclusion Criteria:

* Patients <18 years of age
* Patients who are unable to provide informed consent
* Patients without a positive COVID-19 PCR result obtained through nasopharyngeal swab - Patients with a COVID-19 diagnosis but without self-reported anosmia
* Patients with severe COVID-19 disease as defined by the Mouth Sinai Health System Treatment Guidelines for SARS-COV-2 (requiring high flow nasal cannula, non-rebreather, CPAP/BIPAP, or mechanical ventilation OR patients requiring pressor medication OR patients with evidence of end organ damage)
* Patients with pre-existing self-reported olfactory dysfunction
* Patients with a history of chronic nasal/sinus infections (rhinosinusitis) or history of endoscopic sinus surgery
* Patients using nasal steroid sprays or irrigations for any reason
* Patients who are prisoners of the state
* Patients who have psychiatric or developmental disorder conditions that may impair ability to provide informed consent
* Patients will also be excluded if they have an allergy to fish or an omega-3 supplement, or do not eat fish or fish- containing substances for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred-Marc Iloreta, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaira LA, Salzano G, Deiana G, De Riu G. Anosmia and Ageusia: Common Findings in COVID-19 Patients. Laryngoscope. 2020 Jul;130(7):1787. doi: 10.1002/lary.28692. Epub 2020 Apr 15. PMID 32237238
- [Background] Fonteyn S, Huart C, Deggouj N, Collet S, Eloy P, Rombaux P. Non-sinonasal-related olfactory dysfunction: A cohort of 496 patients. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Apr;131(2):87-91. doi: 10.1016/j.anorl.2013.03.006. Epub 2014 Mar 26. PMID 24679542
- [Background] Hendriks AP. Olfactory dysfunction. Rhinology. 1988 Dec;26(4):229-51. PMID 3070710
- [Background] Eliezer M, Hautefort C, Hamel AL, Verillaud B, Herman P, Houdart E, Eloit C. Sudden and Complete Olfactory Loss of Function as a Possible Symptom of COVID-19. JAMA Otolaryngol Head Neck Surg. 2020 Jul 1;146(7):674-675. doi: 10.1001/jamaoto.2020.0832. No abstract available. PMID 32267483
- [Background] Croy I, Nordin S, Hummel T. Olfactory disorders and quality of life--an updated review. Chem Senses. 2014 Mar;39(3):185-94. doi: 10.1093/chemse/bjt072. Epub 2014 Jan 15. PMID 24429163
- [Background] Reden J, Herting B, Lill K, Kern R, Hummel T. Treatment of postinfectious olfactory disorders with minocycline: a double-blind, placebo-controlled study. Laryngoscope. 2011 Mar;121(3):679-82. doi: 10.1002/lary.21401. Epub 2011 Feb 1. PMID 21287560
- [Background] Vukkadala N, Qian ZJ, Holsinger FC, Patel ZM, Rosenthal E. COVID-19 and the Otolaryngologist: Preliminary Evidence-Based Review. Laryngoscope. 2020 Nov;130(11):2537-2543. doi: 10.1002/lary.28672. Epub 2020 Apr 24. PMID 32219846
- [Background] Ekstrom I, Sjolund S, Nordin S, Nordin Adolfsson A, Adolfsson R, Nilsson LG, Larsson M, Olofsson JK. Smell Loss Predicts Mortality Risk Regardless of Dementia Conversion. J Am Geriatr Soc. 2017 Jun;65(6):1238-1243. doi: 10.1111/jgs.14770. Epub 2017 Mar 22. PMID 28326534
- [Background] Sorokowska A, Drechsler E, Karwowski M, Hummel T. Effects of olfactory training: a meta-analysis. Rhinology. 2017 Mar 1;55(1):17-26. doi: 10.4193/Rhino16.195. PMID 28040824
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Cavazzana A, Larsson M, Munch M, Hahner A, Hummel T. Postinfectious olfactory loss: A retrospective study on 791 patients. Laryngoscope. 2018 Jan;128(1):10-15. doi: 10.1002/lary.26606. Epub 2017 May 29. PMID 28556265
- [Background] Pekala K, Chandra RK, Turner JH. Efficacy of olfactory training in patients with olfactory loss: a systematic review and meta-analysis. Int Forum Allergy Rhinol. 2016 Mar;6(3):299-307. doi: 10.1002/alr.21669. Epub 2015 Dec 1. PMID 26624966
- [Background] Boesveldt S, Postma EM, Boak D, Welge-Luessen A, Schopf V, Mainland JD, Martens J, Ngai J, Duffy VB. Anosmia-A Clinical Review. Chem Senses. 2017 Sep 1;42(7):513-523. doi: 10.1093/chemse/bjx025. PMID 28531300
- [Background] Reden J, Mueller A, Mueller C, Konstantinidis I, Frasnelli J, Landis BN, Hummel T. Recovery of olfactory function following closed head injury or infections of the upper respiratory tract. Arch Otolaryngol Head Neck Surg. 2006 Mar;132(3):265-9. doi: 10.1001/archotol.132.3.265. PMID 16549746
- [Background] Damm M, Pikart LK, Reimann H, Burkert S, Goktas O, Haxel B, Frey S, Charalampakis I, Beule A, Renner B, Hummel T, Huttenbrink KB. Olfactory training is helpful in postinfectious olfactory loss: a randomized, controlled, multicenter study. Laryngoscope. 2014 Apr;124(4):826-31. doi: 10.1002/lary.24340. Epub 2013 Sep 19. PMID 23929687
- [Derived] Lerner D, Garvey K, Arrighi-Allisan A, Filimonov A, Filip P, Liu K, Ninan S, Schaberg M, Colley P, Del Signore A, Govindaraj S, Iloreta AM. Letter to the editor: Study Summary - Randomized Control Trial of Omega-3 Fatty Acid Supplementation for the Treatment of COVID-19 Related Olfactory Dysfunction. Trials. 2020 Nov 23;21(1):942. doi: 10.1186/s13063-020-04905-y. PMID 33225989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with laboratory-confirmed or clinically-suspected COVID-19 infection and self-reported new-onset OD from August 2020 to November 2021 were prospectively recruited from otolaryngology and primary care practices across a large metropolitan health system as well as through a web-based symptom-tracking application and self-referral, resulting in a cohort of individuals from throughout the United States.
Groups:
- Omega-3: 2,000mg daily of O3FA supplementation in the form of 2 capsules of Nature Made® Ultra Omega-3 Fish Oil 1400mg, each of which contains 1000 mg of O3FAs
- Placebo/Control: received a placebo pill of identical size and shape to be taken twice daily.
Period: Overall Study
Arm/Group | Omega-3 | Placebo/Control
Started | 70 | 69
Completed | 57 | 60
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 | Placebo/Control | Total
Number analyzed (Participants) | 57 | 60 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (14.6) | 40.7 (12.7) | 41.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 11 | 14 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Olfactory Dysfunction [Count of Participants; unit: Participants]
  Anosmia | 45 | 47 | 92
  Hyposmia | 4 | 6 | 10
  Parosmia | 1 | 0 | 1
  Hyposmia & Parosmia | 7 | 7 | 14
Anosmia Severity (Worst) [Mean (Standard Deviation); unit: units on a scale] — Full range from 1-100, with higher score indicating more severe
  units on a scale | 91.9 (16.9) | 96.0 (8.54) | 93.9 (13.3)
Anosmia Severity (Current) [Mean (Standard Deviation); unit: units on a scale] — Full range from 1-100, with higher score indicating more severe
  units on a scale | 68.1 (27.7) | 73.2 (22.2) | 70.8 (25.0)
Comorbidities, n (%) [Count of Participants; unit: Participants]
  Ageusia | 41 | 48 | 89
  History of Facial Trauma | 2 | 0 | 2
  Chronic Rhinosinusitis | 1 | 1 | 2
  Allergic Rhinitis | 3 | 6 | 9
  Neurodegenerative Disease | 1 | 0 | 1
Duration of Olfactory Dysfunction Prior to Trial Start [Mean (Standard Deviation); unit: days] | 196 (105) | 204 (95.6) | 200 (99.6)
Therapies Used Prior to Trial Start [Count of Participants; unit: Participants]
  Smell Training | 24 | 24 | 48
  Nasal Saline Spray or Irrigation | 11 | 11 | 22
  Intranasal Corticosteroid Spray or Irrigation | 5 | 5 | 10
  Oral Corticosteroids | 0 | 3 | 3
  Other | 3 | 8 | 11
Concomitant Therapies Used During the Trial, n (%) *** [Count of Participants; unit: Participants]
  Smell Training | 12 | 17 | 29
  Nasal Saline | 5 | 8 | 13
  Intranasal Corticosteroid Spray or Irrigation | 6 | 7 | 13
  Oral Corticosteroids | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Smell Identification Test (BSIT)
Description: Change in BSIT. Brief Smell Identification Test (BSIT) is a 12-item instrument, full range score from 0 to 12, higher score indicates better olfactory performances.
Time Frame: Week 0 and Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 57 | 60
score on a scale
  Baseline | 6.77 (1.94) | 7.20 (1.88)
  Week 6 | 7.89 (2.00) | 7.88 (2.19)
  Change | 1.12 (1.99) | 0.68 (1.86)

2. Primary Outcome: Change in Brief Smell Identification Test (BSIT) in Participants With Severe Olfactory Dysfunction
Description: Mean change in BSIT in participants with severe olfactory dysfunction defined as BSIT ≤ 7. Brief Smell Identification Test (BSIT) is a 12-item instrument, full range score from 0 to 12, higher score indicates better olfactory performances.
Time Frame: Week 0 and Week 6
Population: Participants with severe olfactory dysfunction defined as BSIT ≤ 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 23 | 16
score on a scale | 2.30 (1.77) | 1.63 (1.82)

3. Primary Outcome: Change in Brief Smell Identification Test (BSIT) in Participants With Laboratory-Confirmed COVID-19 and Severe Olfactory Dysfunction
Description: Mean change in BSIT in participants with laboratory-confirmed COVID-19. Brief Smell Identification Test (BSIT) is a 12-item instrument, full range score from 0 to 12, higher score indicates better olfactory performances.
Time Frame: Week 0 and Week 6
Population: Participants with Laboratory-Confirmed COVID-19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 51 | 51
score on a scale | 1.18 (1.88) | 0.61 (1.87)

4. Primary Outcome: Change in Brief Smell Identification Test (BSIT) in Participants With Laboratory-Confirmed COVID-19
Description: Mean change in BSIT in participants with severe olfactory dysfunction defined as BSIT ≤ 6. Brief Smell Identification Test (BSIT) is a 12-item instrument, full range score from 0 to 12, higher score indicates better olfactory performances.
Time Frame: Week 0 and Week 6
Population: Data not collected
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Modified Brief Questionnaire of Olfactory Dysfunction (mQOD-NS)
Description: The modified Brief Questionnaire of Olfactory Dysfunction - Negative Statements (QOD-NS) survey is a 17-item instrument, each item graded on a scale from 0 to 3, with total scale range from 0 to 51. Higher score indicates better olfactory-specific quality of life (QOL).
Time Frame: baseline, weeks 1, 2, 4 and 6 after softgel initiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 57 | 60
score on a scale
  baseline | 12.29 (4.46) | 13.73 (4.33)
  week 1 | 11.41 (4.42) | 12.54 (4.83)
  week 2 | 11.46 (4.81) | 12.76 (4.41)
  week 4 | 11.17 (5.15) | 12.95 (4.67)
  week 6 | 11.19 (4.58) | 12.33 (4.80)

6. Secondary Outcome: Sinonasal Outcomes Test (SNOT-22)
Description: Sino-Nasal Outcome Test (SNOT-22) is a 22-item instrument, total scale range from 0 to 110, higher score indicates more severe QOL impact.
Time Frame: baseline, weeks 1, 2, 4 and 6 after softgel initiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Omega-3 | Placebo/Control
Number analyzed (Participants) | 57 | 60
score on a scale
  baseline | 22.35 (13.23) | 25.75 (12.43)
  week 1 | 21.23 (13.60) | 24.54 (12.90)
  week 2 | 21.41 (14.33) | 22.90 (12.58)
  week 4 | 20.79 (13.56) | 23.47 (13.82)
  week 6 | 19.91 (13.05) | 22.41 (13.58)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Omega-3 | Placebo/Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/69
Other Adverse Events (participants affected / at risk) | 0/70 | 5/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 (N=70) | Placebo/Control (N=69)
worsening of gastroesophageal reflux symptoms (Gastrointestinal disorders) | 0 | 3
unable to swallow the capsules (General disorders) | 0 | 1
Unrelated upcoming surgery (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT04495816/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT04495816/SAP_001.pdf